CLINICAL TRIAL: NCT07066306
Title: Evaluation of the Intraoperative and Postoperative Effects of Local Ketamine Injection in Orthognathic Surgery
Brief Title: Effects of Local Ketamine in Orthognathic Procedures
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E-54022451
Record Dates: First submitted 2025-06-23; First posted 2025-07-15 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Dentofacial Deformities; Analgesia; Vomiting, Postoperative; Nausea, Postoperative
Keywords: orthognthic surgery; ketamine; analgesia; nausea and vomiting
MeSH Terms: conditions — Dentofacial Deformities; Agnosia; Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Ketamine; Carticaine; Epinephrine; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- local ketamine group (Experimental): Following induction of general anesthesia, 0.2 mg/kg of ketamine will be locally administered in place of standard local anesthetic in this group
  Interventions: Drug: Ketamine
- control group (Active Comparator): Following induction of general anesthesia, standard local anesthetic (articaine) will be locally administered in this group
  Interventions: Drug: Articaine Hydrochloride + Epinephrine

INTERVENTIONS:
Drug: Ketamine — In the ketamine group, 0.2 mg/kg of ketamine will be administered locally. This application will be performed twice: once during the Le Fort I osteotomy and once during the sagittal split osteotomy. After calculating the total dose, it will be equally divided and administered locally to both the maxilla and the mandible.
  Arms: local ketamine group
Drug: Articaine Hydrochloride + Epinephrine — A total of 4 ampoules of articaine hydrochloride will be used. Two ampoules will be administered prior to the incision during the Le Fort I osteotomy, and the remaining two ampoules will be used prior to the incision during the sagittal split osteotomy.
  Other Names: local anesthetic
  Arms: control group

SUMMARY:
Orthognathic surgery is performed to correct congenital, developmental, or trauma-related skeletal deformities of the maxilla and mandible. These procedures involve multiple incisions, dissections, and osteotomies, leading to significant postoperative inflammatory responses and acute pain. Postoperative pain is a key factor influencing recovery, return to function, and length of hospital stay.

Various analgesics have been used to manage pain after orthognathic surgery, including NSAIDs, opioids, acetaminophen, NMDA receptor antagonists, and long-acting local anesthetics. Ketamine is a well-known NMDA receptor antagonist with both central and peripheral analgesic effects. In subnesthetic doses, ketamine has been evaluated in various surgical fields for its potential to enhance analgesia when combined with local anesthetics, while minimizing systemic side effects.

Studies have shown that local ketamine administration during cleft palate repair and third molar extractions can significantly reduce postoperative pain, swelling, and trismus. However, to date, no studies have investigated the effects of locally administered ketamine in orthognathic surgery. Therefore, this study was designed to evaluate the intraoperative and postoperative effects of local ketamine injection in this context.

DETAILED DESCRIPTION:
Orthognathic surgery is performed to correct congenital or developmental anomalies of the maxilla and mandible, as well as secondary deformities caused by trauma. These procedures require multiple incisions, dissections, and osteotomies in both the maxilla and mandible. The acute postoperative pain that follows orthognathic surgery is primarily the result of these surgical traumas and the subsequent inflammatory process. As tissue healing progresses, postoperative pain gradually subsides. This type of pain is one of the primary factors affecting postoperative recovery, return to function, and length of hospital stay.

Many studies have focused on achieving optimal analgesia during this period, which significantly affects patients' postoperative quality of life. For this purpose, several agents have been used, including non-steroidal anti-inflammatory drugs (NSAIDs), opioids, non-opioid analgesics (such as acetaminophen), NMDA receptor antagonists, and long-acting local anesthetics.

Ketamine is a well-known general anesthetic and short-acting intraoperative analgesic agent with established pharmacodynamic and pharmacokinetic profiles and known side effects. Ketamine is a non-selective antagonist of supraspinal N-methyl-D-aspartate (NMDA) receptors. It is believed that inhibition of these receptors reduces neuronal excitation and produces analgesia through this mechanism. Ketamine's interactions with spinal pain receptors and opioid receptors are also thought to contribute to its analgesic effects.

In low doses, ketamine has been evaluated for local analgesic purposes in combination with local anesthetics in various surgical procedures, aiming to minimize side effects. Cleft palate repair and third molar extractions are among the oral surgery procedures where the local analgesic efficacy of ketamine has been investigated. In a study by Jha et al. on cleft palate repair, the authors examined the effects of local bupivacaine combined with ketamine on postoperative nausea, vomiting, dysphagia, and sleep patterns. They found that patients in the ketamine group had superior outcomes in terms of reduced need for additional analgesia, improved sleep, and earlier return to feeding.

Similarly, in the literature some studies reported that significant reductions in postoperative pain, swelling, and trismus in third molar extraction patients when sub-anesthetic doses of ketamine were combined with local anesthetics. Shah et al. also observed that combining ketamine with local anesthetics during third molar extraction reduced postoperative pain and swelling compared to local anesthetics alone.

To date, there are no studies in the literature investigating the effects of combining ketamine with local anesthetics in orthognathic surgery. Therefore, this study was designed to address this gap.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Class II or Class III skeletal deformities who underwent bimaxillary orthognathic surgery due to dentofacial deformities.
2. ASA I-II physical status patients.
3. Patients aged between 18 and 45 years.
4. Patients who received anesthesia induction and maintenance with propofol (0.2-0.6 mg/kg/hour) titrated to maintain an entropy score between 40-60, and remifentanil (0.05-0.5 mg/kg/hour) adjusted to maintain a Surgical Pleth Index (SPI) between 20-50.
5. Patients who received a combination of local anesthetic and ketamine.
6. Patients who were administered patient-controlled analgesia (PCA) at the end of the surgery and whose opioid consumption via PCA was monitored during the first 24 hours postoperatively.
7. Patients whose nausea-vomiting scores and need for antiemetics were recorded.
8. Patients with complete documentation of anesthesia records, including entropy scores, SPI values, and total doses of propofol and remifentanil administered.
9. Patients with completed postoperative edema follow-up forms.

Exclusion Criteria:

1. Patients with a known allergy to ketamine.
2. Patients with uncontrolled systemic diseases.
3. Patients using psychotropic medications.
4. Patients with a history of substance abuse.
5. Patients with chronic pain lasting longer than 3 months.
6. Patients using analgesic or hypnotic medications for more than 2 weeks.
7. Cases in which complications occurred during surgery that required deviation from the standard orthognathic surgical protocol and could potentially affect postoperative pain levels (e.g., bad split, unexpectedly prolonged surgical duration, etc.).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-21 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
rescue analgesia dose | 2 days
  In the postoperative period, in addition to the standard pain management protocol, the need for rescue analgesia will be recorded by calculating the total administered dose. For rescue analgesia, 50 mg of tramadol will be delivered via infusion pump and administered through patient-controlled analgesia (PCA).
postoperative edema calculation for the first 1-3 and 7 day (cm) | 7 days
  the first secondary outcome of this study is post operative edema: Prior to anesthesia induction, Tragus (Tra) and Gonion (Go) points were marked with methylene blue, and distances including Lateral Canthus - Gonion, Tragus-Commissure, and interincisal distances were measured with a paper ruler and recorded as preoperative measurements.Measurements of Lateral Canthus - Gonion, Tragus-Commissure, and Interincisal distances were repeated on postoperative days 1, 3, and 7 for evaluating postoperative edema.
Visual analogue scale | 2 days
  Author asses the pain score with visual analogue scale (VAS) every 2 hours interval with 2. days. Higher scores means patients feel more pain and lower scores mean patients feel low pain. minımum score is 0, and maximum is 100.

SECONDARY OUTCOMES:
nausea and vomiting | 3 days
  after the operation investigator assess the nausea and vomiting every 2 hours interval and score it in 4 point scale
  Nausea and Vomiting Scoring System:
  0 = No nausea
  1. = Nausea only
  2. = Nausea accompanied by retching
  3. = Vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf Universty, Istanbul, Fatih, Turkey (Türkiye)